CLINICAL TRIAL: NCT01198405
Title: A Prospective,Randomized,Open-labeled,and Blind Endpoint Study of Enhanced External Counterpulsation for Patients With Coronary Heart Disease
Brief Title: Study of Enahnced External Counterpulsation to Treat Coronary Heart Disease
Acronym: PROBE-EECP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Gui-Fu Wu, The First Affiliated Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSU-5010-2008
Record Dates: First submitted 2010-07-29; First posted 2010-09-10 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; enhanced external counterpulsation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced External Counterpulsation (Experimental): Treatment of Enhanced External Counterpulsation (EECP) with a prespecified protocol on top of guideline-driven standard medical therapy.
  Interventions: Device: Enhanced external counterpulsation
- Control (Active Comparator): Guideline-driven standard medical therapy.
  Interventions: Drug: Guideline-driven standard medical therapy

INTERVENTIONS:
Device: Enhanced external counterpulsation — Treatment of enhanced external counterpulsation (EECP) with a prespecified protocol on top of a guideline-driven standard medical therapy. EECP Protocol is defined as a standard session of a total of 36 hours of EECP treatment, given one hour per day, six days per week. The same session is thereafter repeated at least once every year.
  Arms: Enhanced External Counterpulsation
Drug: Guideline-driven standard medical therapy — Standard management, both pharmacological and non-pharmacological, given according to current practice guidelines at the discretion of clinicians
  Arms: Control

SUMMARY:
To investigate the mid- and long-term effect of Enhanced External Counterpulsation combined with guideline-driven standard treatment on patients documented with and/or at high risk of coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* at least one coronary lesion of more than 50% stenosis shown by angiography
* history of acute myocardial infarction(at least one month before)
* history of prior revascularization (Percutaneous Coronary Intervention or Coronary Artery Bypass Grafting)
* typical angina episodes with evidence of myocardial ischemia
* Signed informed consent

Exclusion Criteria:

* Obvious aortic insufficiency, aortic aneurysm, aortic dissection
* Coronary fistula or severe coronary aneurysm
* Symptomatic Congestive heart failure
* Valvular heart disease, congenital heart diseases, cardiomyopathies
* Cerebral hemorrhage within six months, bleeding disorders or identified bleeding tendency;
* Lower limb infection, phlebitis, varicosity, deep venous thrombosis;
* Progressive malignancies or diseases with poor prognosis;
* uncontrolled hypertension, defined as SBP≥180mmHg or DBP≥110mmHg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
composite endpoint of rate of all-cause mortality, revascularization, rehospitalization and acute myocardial infarction | up to 5 years

SECONDARY OUTCOMES:
vascular endothelial function | up to 5 years
  measurment of flexibility of peripheral artery and flow-mediated dilatation (FMD)
cardiac structure and exercise tolerance | up to 5 years
  cardiac chamber diameter, left ventricular wall thickness, ejection fraction, and etc., as deternmined by echocardiographic examination; exercise tolerance, as determined by Treadmill's Test
new-onset diabetes | up to 5 years
  fasting, postprandial and random plasma glucose levels; glycosylated hemoglobin A1c (GHbA1c)
atherosclerosis | up to 5 years
  peripheral artery: plaque of common carotid artery, carotid intima-media Thickness, systolic and diastolic blood pressure (SBP & DBP)
24-hour urinary protein | up to 5 years
  24-hour urinary protein/albumin by urinalysis
all-cause mortality | up to 5 years
revascularization rate | up to 5 years
rehospitalization rate | up to 5 years
rate of acute myocardial infarction | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-min Du, M.D., Principal Investigator — The 1st Affiliated Hospital of Sun Yat-sen University; Gui-fu Wu, M.D. & Ph.D., Study Director — The 1st Affiliated Hospital of Sun Yat-sen University
Locations (4):
- China (4):
  - The 1st Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The 2nd Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The 3rd Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The 5th Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong

REFERENCES:
- [Background] Loh PH, Cleland JG, Louis AA, Kennard ED, Cook JF, Caplin JL, Barsness GW, Lawson WE, Soran OZ, Michaels AD. Enhanced external counterpulsation in the treatment of chronic refractory angina: a long-term follow-up outcome from the International Enhanced External Counterpulsation Patient Registry. Clin Cardiol. 2008 Apr;31(4):159-64. doi: 10.1002/clc.20117. PMID 18404725
- [Background] Kitsou V, Xanthos T, Roberts R, Karlis GM, Padadimitriou L. Enhanced external counterpulsation: mechanisms of action and clinical applications. Acta Cardiol. 2010 Apr;65(2):239-47. doi: 10.2143/AC.65.2.2047060. PMID 20458834
- [Background] Manchanda A, Soran O. Enhanced external counterpulsation and future directions: step beyond medical management for patients with angina and heart failure. J Am Coll Cardiol. 2007 Oct 16;50(16):1523-31. doi: 10.1016/j.jacc.2007.07.024. Epub 2007 Oct 1. PMID 17936150
- [Background] Michaels AD, McCullough PA, Soran OZ, Lawson WE, Barsness GW, Henry TD, Linnemeier G, Ochoa A, Kelsey SF, Kennard ED. Primer: practical approach to the selection of patients for and application of EECP. Nat Clin Pract Cardiovasc Med. 2006 Nov;3(11):623-32. doi: 10.1038/ncpcardio0691. PMID 17063167
- [Background] Cohn PF. Enhanced external counterpulsation for the treatment of angina pectoris. Prog Cardiovasc Dis. 2006 Sep-Oct;49(2):88-97. doi: 10.1016/j.pcad.2006.04.001. PMID 17046434
- [Background] O'Rourke MF, Hashimoto J. Enhanced external counterpulsation why the benefit? J Am Coll Cardiol. 2006 Sep 19;48(6):1215-6. doi: 10.1016/j.jacc.2006.06.036. Epub 2006 Aug 28. No abstract available. PMID 16979008
- [Background] Michaels AD, Raisinghani A, Soran O, de Lame PA, Lemaire ML, Kligfield P, Watson DD, Conti CR, Beller G. The effects of enhanced external counterpulsation on myocardial perfusion in patients with stable angina: a multicenter radionuclide study. Am Heart J. 2005 Nov;150(5):1066-73. doi: 10.1016/j.ahj.2005.01.054. PMID 16291000
- [Background] Arora RR, Chou TM, Jain D, Fleishman B, Crawford L, McKiernan T, Nesto R, Ferrans CE, Keller S. Effects of enhanced external counterpulsation on Health-Related Quality of Life continue 12 months after treatment: a substudy of the Multicenter Study of Enhanced External Counterpulsation. J Investig Med. 2002 Jan;50(1):25-32. doi: 10.2310/6650.2002.33514. PMID 11813825
- [Background] Arora RR, Chou TM, Jain D, Fleishman B, Crawford L, McKiernan T, Nesto RW. The multicenter study of enhanced external counterpulsation (MUST-EECP): effect of EECP on exercise-induced myocardial ischemia and anginal episodes. J Am Coll Cardiol. 1999 Jun;33(7):1833-40. doi: 10.1016/s0735-1097(99)00140-0. PMID 10362181